CLINICAL TRIAL: NCT03905291
Title: A Randomized, Double-blinded, Placebo-controlled, Single Center, Dose Escalation, Phase I Study to Evaluate the Pharmacokinetic/Pharmacodynamic Characteristics and Safety/Tolerability of MT921 in Healthy Subjects
Brief Title: Pharmacokinetic/Pharmacodynamic Characteristics and Safety/Tolerability of MT921 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT11-KR17SMF115
Record Dates: First submitted 2019-03-25; First posted 2019-04-05 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MT921 60mg Group (Experimental): MT921 60 mg
  Interventions: Drug: MT921
- MT921 120mg Group (Experimental): MT921 120 mg
  Interventions: Drug: MT921
- MT921 150mg Group (Experimental): MT921 150 mg
  Interventions: Drug: MT921
- Placebo Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT921 — Formulated as an injectable solution
  Arms: MT921 120mg Group; MT921 150mg Group; MT921 60mg Group
Drug: Placebo — normal saline
  Arms: Placebo Group

SUMMARY:
To determine the pharmacokinetic/pharmacodynamic characteristics and safety/tolerability of MT921 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 20 and 65 years

Exclusion Criteria:

* Subject not appropriate for participating in this study according to the investigator's opinion

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) measured by Liquid Chromatography-mass spectrometry (LC/MS) | Up to 24 hours
  Peak plasma concentration measured by Liquid Chromatography-mass spectrometry (LC/MS) achieving in the test area of the body after administration.
AUC0-24 | Up to 24 hours
  Area under the plasma concentration versus time curve from time 0 to 24 hours measured by Liquid Chromatography-mass spectrometry (LC/MS) after administration
Maximum Time (Tmax) measured by Liquid Chromatography-mass spectrometry (LC/MS) | Up to 24 hours
  The time at which the Cmax is observed measured by Liquid Chromatography-mass spectrometry (LC/MS).
Half-life (t1/2) measured by Liquid Chromatography-mass spectrometry (LC/MS) | Up to 24 hours
  The time it takes for the concentration of the drug in the plasma or the total amount in the body to be reduced by 50% measured by Liquid Chromatography-mass spectrometry (LC/MS).

OTHER OUTCOMES:
Number of participants with adverse events as assessed by MedDRA version 17.0 | Up to 21 days
  Assessment of safety in investigational product with the number of participants with adverse events as assessed by MedDRA version 17.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Anam Hospital, Seoul, South Korea